CLINICAL TRIAL: NCT04577248
Title: The Prospecive OBSERVational Munich Interventional MITRAl-Valve Registry
Acronym: OBSERV-MITRA
Status: Recruiting | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GE DHM-AN-EHK-2020/09
Record Dates: First submitted 2020-10-01; First posted 2020-10-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Mitral Valve Regurgitation; Mitral Valve Stenosis; Tricuspid Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Stenosis; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: edge-to-edge valve repair — edge-to-edge valve repair

SUMMARY:
Prospective, single-center observational registry including all consecutive patients treated with transcatheter mitral or tricuspid valve therapy at the Deutsches Herzzentrum München, Germany.

DETAILED DESCRIPTION:
Long-term mortality after transcatheter mitral or tricuspid valve therapy

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years and consentable
* Mitral Valve Regurgitation, Mitral Valve Stenosis, Tricuspid Valve Regurgitation, Tricuspid Stenosis
* Transcatheter mitral or tricuspid valve therapy considered best option by heart-team decision
* Written informed consent

Exclusion Criteria:

* Patient's inability to fully cooperate with the protocol

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population treated with transcatheter mitral or tricuspid valve therapy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Long-term mortality | 5 years
  Long-term mortality

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mayr, MD, Study Chair — Dept. of Anesthesiology, Deutsches Herzzentrum München; Michael Joner, Prof, Study Chair — Dept. of Cardiology, Deutsches Herzzentrum München; Tobias Rheude, MD, Principal Investigator — Dept. of Cardiology, Deutsches Herzzentrum München; Costanza Pellegrini, MD, Principal Investigator — Dept. of Cardiology, Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München des Freistaates Bayern, Technische Universität München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No